CLINICAL TRIAL: NCT02344537
Title: Meditation and Stretching for Post Treatment Lyme Disease Syndrome
Acronym: LMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We aimed for 40, but slow enrollment and limited funds led us to terminate the study before completing full enrollment
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Psychiatry, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6927
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2022-11

CONDITIONS: Post Treatment Lyme Disease Syndrome
Keywords: Lyme DIsease; Kundalini Yoga
MeSH Terms: conditions — Post-Lyme Disease Syndrome; Lyme Disease | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meditation Group Therapy (Experimental): Kundalini Yoga incorporates mindfulness practice with a triad of stretching, breathing, and meditation. The three components of treatment consist of muscular relaxation/stretching exercises, a meditation period characterized by a directed breathing exercise, and then a guided meditation.
  Interventions: Behavioral: Kundalini Yoga
- Wait-List Controls (No Intervention): The wait-list group will not take part in study treatment (daily meditation or stretching) during the study wait of 8 weeks in order for us to compare change related to the study intervention to change associated with no active treatment ( treatment-as-usual). (After completing 8 weeks of no study treatment as part of the wait-list group, these patients will be offered the opportunity to receive 8 weeks of treatment.)

INTERVENTIONS:
Behavioral: Kundalini Yoga — Kundalini Yoga incorporates mindfulness practice with a triad of stretching, breathing, and meditation. The three components of treatment consist of muscular relaxation/stretching exercises, a meditation period characterized by a directed breathing exercise, and then a guided meditation.
  Other Names: Relaxation, stretching and meditation
  Arms: Meditation Group Therapy

SUMMARY:
The investigators wish to conduct a preliminary study to examine the efficacy of meditation among patients with Post Treatment Lyme Syndrome (PTLDS). Specifically, the investigators will use the breathing, meditation, and stretching techniques common to Kundalini Yoga practice. The investigators plan to assess the degree in which this practice can reduce Post-Treatment Lyme Disease symptoms. Because fatigue and pain are so common among patients with PTLDS, the primary focus of this study will be fatigue and pain. Secondary outcomes will include cognitive complaints, physical and mental functioning, medical utilization, somatic symptoms, and psychopathology.

DETAILED DESCRIPTION:
The CDC reports that approximately 10-20% of patients treated for Lyme disease with the IDSA-recommended 2-4 week course of antibiotics will continue to have symptoms of fatigue, pain, or joint and muscle aches despite prior antibiotic treatment. The symptoms can last months or even years after treatment. The medical community officially calls this condition "Post-treatment Lyme disease Syndrome" (PTLDS) but some have called it "chronic Lyme disease." Because some patients with PTLDS continue to have ongoing symptoms despite many additional courses of antibiotics beyond the standard course, alternative non-antibiotic treatment programs need to be explored. The proposed study seeks to evaluate the efficacy of meditation among those patients that have been previously treated for Lyme disease but are still continuing to experience prominent symptoms of fatigue and/or pain.

During this study, patients will be screened initially over the telephone to assess eligibility, sign consent with the study treating psychiatrist, and complete self-report questionnaires. Forty patients will be enrolled. Of these, 20 will be randomly assigned to meditation group therapy and 20 will be assigned to a wait-list. Assessments will be conducted prior to treatment, at 4 weeks and at 8 weeks. There will also be a 6 month follow-up by questionnaire and telephone interview. Study participants randomized to the wait-list control group will then be offered, after 8 weeks, the option of joining a meditation group for 8 weeks. Each meditation group will be composed of 6-8 subjects.

Should this study find evidence suggesting that meditation therapy is helpful in reducing the symptoms of PTLDS, this would be a valuable finding that would lead to a larger study as it has important public health implications for many individuals now quite disabled with these chronic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* History of prior diagnosis of Lyme Disease at least 6 months prior to assessment

  1. EM Rash seen by health professional

     -OR-
  2. History of physician diagnosed disseminated Lyme disease
* Previously treated for Lyme Disease with antibiotics appropriate for stage of disease
* Current symptoms of PTLDS started within 6 months after getting Lyme disease
* Current symptoms have been present for at least the last 6 months.
* Between the ages of 18 and 65, English speaking, male or female
* Primary complaint of fatigue or pain meeting predetermined severity criteria
* Individuals whose medical and/or psychiatric treatment has been stable for the prior 8 weeks
* Individuals who agree to not start a new treatment for PTLS during the course of the study; this applies to both those assigned to the control wait list group and those assigned to the experimental group.

Exclusion Criteria:

* Individual with another reasonable medical explanation (other than Lyme) that might better account for current fatigue or pain (e.g., Thyroid Disease, Anemia, Rheumatoid Arthritis)
* Individual with a major psychiatric diagnosis that might make study participation difficult (e.g, Dissociative Identity Disorder, Psychosis, Post Traumatic Stress Disorder, Substance abuse with the prior 6 months, Pain Disorder treated with opiate-based medication)
* Individuals with severe depression
* Individuals with Physical disability that might make study participation difficult
* Individuals whose current medical status is so severe or unstable that participation in the study (and not receiving new treatments from other providers) would be difficult.
* Unwillingness to complete questionnaires, speak with study research assistant, or dedicate twenty minutes daily to meditation and stretching
* Suicide attempts within the last 6 months or current suicidal thoughts
* Individuals unwilling to delay starting optional treatment for Lyme disease for the duration of the study
* Individuals with a prior lifetime practice of at least one month of daily practice of MBSR or mindfulness or those who currently practice daily meditation or yoga

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Fallon, MD, Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (2):
- United States (2):
  - Private Practice Office of Dr. Alexander, Southport, Connecticut
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Background] Collins C. Yoga: intuition, preventive medicine, and treatment. J Obstet Gynecol Neonatal Nurs. 1998 Sep-Oct;27(5):563-8. doi: 10.1111/j.1552-6909.1998.tb02623.x. PMID 9773368
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] van der Lee ML, Garssen B. Mindfulness-based cognitive therapy reduces chronic cancer-related fatigue: a treatment study. Psychooncology. 2012 Mar;21(3):264-72. doi: 10.1002/pon.1890. Epub 2010 Dec 19. PMID 22383268
- [Background] Grossman P, Kappos L, Gensicke H, D'Souza M, Mohr DC, Penner IK, Steiner C. MS quality of life, depression, and fatigue improve after mindfulness training: a randomized trial. Neurology. 2010 Sep 28;75(13):1141-9. doi: 10.1212/WNL.0b013e3181f4d80d. PMID 20876468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meditation Group Therapy | Wait-List Controls
Started | 16 | 10
Completed | 12 | 8
Not Completed | 4 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Subject started another treatment after wk 6 | 1 | 0
Not completed — Participants completed the treatment but the week 8 data not available. | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meditation Group Therapy | Wait-List Controls | Total
Number analyzed (Participants) | 16 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (13.0) | 62.6 (14.5) | 53.4 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 8 | 21
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Fatigue (Self-reported Level of Fatigue as Measured by the PROMIS Fatigue Scale)
Description: Self-reported assessment of fatigue as measured by the 7 item PROMIS Fatigue Scale. The raw score range is 7-35. The raw score is converted to a T-score with a mean of 50 and a standard deviation of 10; the results reported here are the T-scores. HIgher scores indicate greater fatigue
Time Frame: Assessed at week 4 and 8; week 8 value is reported (primary endpoint). 6 month assessment not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 63.74 (6.46) | 57.15 (9.44)

2. Primary Outcome: Pain Interference (PROMIS Pain Interference Scale)
Description: Self-reported assessment of pain interference as measured by the 6-item PROMIS Pain Interference Scale. The raw score range is 6-30. The raw score is converted to a T-score with a mean of 50 and a standard deviation of 10; the results reported here are the T-scores. HIgher scores indicate greater pain interference.
Time Frame: Assessed at weeks 4 and 8; week 8 data reported (primary endpoint). 6 month assessment not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 61.08 (11.68) | 52.9 (8.28)

3. Primary Outcome: Global Health (Self-reported Levels of Satisfaction With Global Health)
Description: Self-reported assessment of satisfaction with global health as measured by the 1st item ( a 5 point scale, range 1-5) on the PROMIS Global Heath Scale where higher scores indicate greater satisfaction with health.
Time Frame: Assessed at week 4 and 8; week 8 is reported (primary endpoint). 6 month assessment not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 2.58 (1.3) | 2.62 (0.74)

4. Secondary Outcome: Physical Functioning (as Measured by the PROMIS Physical Functioning Scale)
Description: Self-reported assessment of physical functioning as measured by the PROMIS Physical Functioning 8 item Scale. Raw score range 8-40. The raw score is converted to a T-score with a mean of 50 and a standard deviation of 10; the results reported here are the T-scores. HIgher scores indicate better physical functioning.
Time Frame: Assessed at weeks 4 and 8; week 8 data reported (primary endpoint). Month 6 assessment not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 37.41 (8.56) | 41.26 (4.63)

5. Secondary Outcome: General Symptom Questionnaire-30 (Self-reported Symptom Burden)
Description: Self-reported assessment of symptom burden as measured by the 30 item multisystem Global Symptom Questionnaire. Range is 0-120 where higher scores indicate greater symptom burden
Time Frame: Assessed at 4 and 8 weeks; 8 week values are reported (primary endpoint). Month 6 assessment not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 54.9 (26.48) | 29.5 (16.32)

6. Secondary Outcome: Beck Depression Inventory
Description: Self reported mood as measured by the 21 item Beck Depression Inventory. Range is 0-63 where higher scores indicate greater depression.
Time Frame: Assessed at weeks 4 and 8; 8 week data is reported (primary endpoint). Month 6 assessment not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 16 (10.72) | 11 (8.19)

7. Secondary Outcome: PROMIS Social Satisfaction
Description: Assesses satisfaction with social functioning. 8 item scale. Raw score range i 8-40). The raw score is converted to a T-score with a mean of 50 and a standard deviation of 10; the results reported here are the T-scores. HIgher scores indicate greater satisfaction with social functioning.
Time Frame: Assessed at 4 and 8 weeks; 8 week values are reported (primary endpoint). 6 month assessment was not conducted. .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 38.75 (6.85) | 46.56 (5.86)

8. Secondary Outcome: Applied Cognition General Concerns Short-form
Description: This self-report NeuroQoL measure assesses general concerns about cognition. This is an 8 item scale, with raw scores ranging from 8 to 40. The raw score is converted to a T-score with a mean of 50 and a standard deviation of 10; the results reported here are the T-scores. Higher scores mean fewer cognitive concerns.
Time Frame: Assessed and 4 and 8 weeks; the 8 week results are reported (primary outcome timepoint). The 6 month assessment was not conducted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meditation Group Therapy | Wait-List Controls
Number analyzed (Participants) | 12 | 8
score on a scale | 31.66 (7.77) | 37.6 (4.4)

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events over an 8 week period.
Arm/Group | Meditation Group Therapy | Wait-List Controls
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02344537/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT02344537/SAP_001.pdf